CLINICAL TRIAL: NCT02078804
Title: SCREESCO - Screening of Swedish Colons
Brief Title: Colonoscopy and FIT as Colorectal Cancer Screening Test in the Average Risk Population
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University Hospital (Other)
Collaborators: Swedish Association of Local Authorities and Regions (Other)
Responsible Party: Principal Investigator, Anna Forsberg, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: 2012/2058- 31/3
Record Dates: First submitted 2014-02-11; First posted 2014-03-05 (Estimated); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Mortality; Incidence; Screening; Health-economy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Colonoscopy (Experimental): 20 000 subjects will be invited to an once-only colonoscopy.
  Interventions: Procedure: Colonoscopy
- FIT for occult blood (Experimental): 60 000 persons will be invited to take a fecal test for hemoglobin year 1 and year 3. If test-positive, they will be referred to colonoscopy.
  Interventions: Procedure: Colonoscopy
- Controls (No Intervention): 120 000 matched persons will be identified in the Swedish Register of the total population and will be used as controls.

INTERVENTIONS:
Procedure: Colonoscopy — 20 000 individuals will be randomised to a primary screening colonoscopy and 60 000 to take a feces test for occult blood (FIT) and if positive (10% of individuals) they will be offered a follow-up colonoscopy.
  Arms: Colonoscopy; FIT for occult blood

SUMMARY:
Colorectal cancer (CRC) is a major cause of death in Sweden. There are approximately 6000 new cases each year in Sweden and the disease specific mortality is more than 40%. There risk is about 1% to develop CRC between 60-70 years of age making 60-year olds a suitable target population for colorectal cancer screening.

The Swedish ministry of health and social affairs proposed a national study on the efficiency of colorectal cancer screening in the Swedish population regarding mortality, but also what screening method to be used. Eighteen participating counties of Sweden now fund the study to be launched in 2014.

From the Register of the total population individuals 59-62 years of age will be randomized and invited by mail to screening. Thirty- thousand five hundred individuals will be invited to primary colonoscopy and 60 000 individuals will be invited to high sensitive FIT (approximately 10% positive) and if positive to a subsequent follow-up colonoscopy. If test negative a second round of FIT will be asked for in two years. In total 183 000 randomized individuals will not be invited to screening, but followed in the Swedish Cancer register and serve as controls. The inclusion period I set to five years (five years with the second round of FIT) generating approximately 5 000 colonoscopies yearly the first three years and 1200 year four and five at a compliance rate of 35% in the colonoscopy arm and 50% in the FIT arm.

Follow-up time is set to 15 years with the primary endpoint disease specific mortality, but also incidence. Secondary outcomes by others to be studied are in short quality assurance variables of colonoscopy, participants and non-participants experiences of the invitation and the screening procedure, health economy measures of the CRC-screening study and when implemented in clinical care.

DETAILED DESCRIPTION:
Background: The primary purpose of cancer screening is to reduce mortality from the disease in the population by finding the cancer at an early and treatable stage. The cancer has to be an important health problem to be a suitable target for screening. With approximately 6 000 new cases each year in Sweden (Cancer register), colorectal cancer (CRC) is the third most common cancer in Sweden and the five-year survival rate is close to 60%, but when detected at an early stage the rate is 90%.

Both larger precursor stages - the adenomatous polyp (Muto, Vogelstein) - and cancers could be detected by sensitive methods to analyze blood in the stool. Removal of adenomas has a protective effect against colorectal cancer development (Winawer, Muller, Thiis-Evensen) and, consequentially, a colorectal cancer screening program also have the potential of decreasing the future incidence of the disease.

The screening test must be free from unwanted side effects, inexpensive, but also simple to take and easy to interpret (Armitage). Furthermore, a high sensitivity and specificity is a prerequisite for a screening test to be used in a program of the average risk population.

Indirect tests: The most commonly used screening test has been the guaiac based fecal occult blood test (Hemoccult®). Four larger RCTs have demonstrated a 16% decreased in CRC mortality with the test in screening (Mandel, Kronborg, Hardcastle, Lindholm). More advanced fecal immunological tests (FITs) with higher sensitivity, but only a marginally increase in specificity, are now available. FIT demonstrates presence of human blood only and no dietary restrictions are needed.

Direct tests: The main advantages with endoscopy are the direct visualization of the colorectum and the possibility of obtaining tissue samples from suspected cancer lesions for histopathology and removing adenomatous polyps. Recently, three RCTs with sigmoidoscopy as the primary screening test have demonstrated both a reduced disease specific mortality of around 30%, but also a reduced incidence of CRC of as much as 40% (Atkin, Segnan, Schoen).

Up to now, there are no larger randomized controlled studies of the average risk population published demonstrating a disease specific mortality reduction with colonoscopy as the primary screening test.

Compliance: compliance is the proportion of individuals offered a screening test and actually take the test (Armitage). The compliance to a screening program is a major determinant of the programs effectiveness - only those who participate can contribute to the mortality reduction achieved by the screening program and with low participation the number of deaths prevented will be few.

A call for a Swedish study of colorectal cancer screening: The Swedish minister of Health and Social affairs, Göran Hägglund, funded a task force in 2011 in order to design a study of the effectiveness of colorectal cancer screening of the average risk population of Sweden. The present study was designed based on what data was needed to get better outcome of colorectal cancer screening in Sweden. All counties participate except for Stockholm and Gotland, due to the already implemented CRC-screening program with Hemoccult®, and the county of Västernorrland.

Material and Methods - study population: In total 200 000 individuals and residents of Sweden will be randomized from the Register of the total population (Register of the total population). The randomized individuals will turn 60-years old the calendar year of randomization. Thirty thousand five hundred individuals will be invited to a primary screening colonoscopy, 60 000 individuals will be invited to high sensitive FIT and, if positive, to a subsequent colonoscopy and 183 000 persons will serve as controls. The inclusion period is set to five years with a repeated test after two years in the FIT arm.

Invitation procedures - FIT: All individuals randomized to FIT as primary screening test will by regular mail receive an invitation to participate in the study. The invitation includes a brochure with information about the incentives of the study and the need for a follow-up colonoscopy in case of a positive test. The invitation contains a FIT-kit for two separate test samples and instructions on how to take the test. With the invitation is a pre-paid return-envelope.

Colonoscopy: All individuals randomized to the colonoscopy arm will receive an invitational letter by regular mail including the brochure with information about the incentives of the study. The invitee will be informed that they shortly by mail will receive an appointment for colonoscopy, sent from the endoscopy clinic in their area of residency.

Controls: The individuals randomized to the control arm will not be contacted and informed about participation as controls in the study. If any individuals would contact the Head secretariat to ask about if they are controls, information will be given.

Interventions - FIT-arm: We plan two rounds of FIT, one the first year and one the third year. We will follow the findings and perform interim analyses and suggest that further rounds of FIT are carried out if the scientific committee deems it necessary. Two tests per round will be asked for without dietary restrictions. If 50% of the invitees comply and send their FIT test to the laboratory (experiences from the ongoing screening program in the counties of Stockholm and Gotland) and 10% are positive, this will generate approximately 1 200 colonoscopies for each year in the FIT-arm except for year four when the number of generated colonoscopies is estimated to 2 400 due to the second round re-testing.

Colonoscopy-arm: A primary screening colonoscopy will be carried out once and with an estimated adherence of about 35%, approximately 10 000 colonoscopies will be carried out. The examination will be performed with or without sedation following a standard bowel cleaning preparation. The endoscopy centers will be accredited and the quality of the examiners will be investigated. The preparations of the bowel will be standardized. All details will follow the European guidelines (von Karsa, Rembacken).

There will be a thorough evaluation of each endoscopist from a quality aspect according to set guidelines. This will be carried out by using a specific quality register in the IT-system where data on the success rate of the colonoscopist, findings and side effects will be entered from all the estimated 17 000 colonoscopies. In the study registry, adverse advents such as pain, bleeding and perforations will also be collected. The register data will continuously be cross-linked with data from the National Patient register (Patient register) and the Swedish Causes of Death register (Cause of death register) in order to find severe adverse events.

Follow-up: Follow-up time is set at 15 years after inclusion and invitation for the primary endpoints colorectal cancer mortality and incidence with interim analysis at 5 and 10 years. Data of all 200.000 individuals randomized from the population register will be obtained from the Causes of Death register (19) and the Cancer register (1). Regarding secondary outcomes, information will be retrieved from other national registries such as the Patient register (18).

Ethical considerations: The study has been processed and approved by the regional Ethics Review Board at Karolinska Institutet, Stockholm, Sweden (No. 2012/2058-31/3).

Statistical analyses: The lifetime cumulative mortality in colorectal cancer in Sweden is about 1% after 15 years. With a 80% power and a 2.5% significance level according to the Bonferroni method the present study need to randomize 30 500 persons in the colonoscopy arm, 60 186 in the FIT arm and 183 372 in the control arm. Based on previous studies, we estimate that the reduction in mortality to about 30% for those examined with FIT and a subsequent colonoscopy and approximately 35% for individuals who are examined with a primary colonoscopy. The compliance is estimated to about 50% in the FIT-arm and approximately 10% of them will have a positive test and invited to follow-up colonoscopy with 80-90% adherence rate. Compliance with primary colonoscopy is estimated to 50% and there is supposed to be a very low contamination from opportunistic screening.

ELIGIBILITY:
Inclusion Criteria:

* People 59-62 years old living in Sweden randomized and identified through the Register of the total population.

Exclusion Criteria:

* Residents of the counties of Stockholm, Gotland and Västernorrland, individuals with diagnosed with colorectal cancer and/or anal cancer, and individuals randomized to be included in the ongoing NordICC-trial.

Ages: 59 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 278000 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality from colorectal cancer in the Swedish population. | 15 years follow-up

SECONDARY OUTCOMES:
Incidence of colorectal cancer in the Swedish population. | 15 years follow-up
To study compliance with the screening program (read study) and what factors are of importance for the adherence rate. | 1-5 years
To study health economy and costs for colorectal cancer screening. | 1-20 years
To study the emotional impact of screening on participants and non-participants including eventual change in lifestyle after invitation and/or participation. | 1-5 years
To study quality control aspects and side effects of screening with colonoscopy. | 1-5 years
To study pathology by means of quality registries and digital pathology. | 1-5 years
To study surveillance strategies for adenomas found at colonoscopy. | 1-20 years
To study associations of DNA in blood with findings at colonoscopy. | 1-20 years
To study the flora of fecal bacteria among participants and outcome of FIT and colonoscopy. | 1-5 years

CONTACTS AND LOCATIONS:
Overall Officials: Anna Forsberg, MD PhD, Principal Investigator — Karolinska Institutet

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cancer register: http://www.socialstyrelsen.se/register/halsodataregister/cancerregistret/inenglish: National Board of Health and Welfare; [cited 2014 February].
- [Background] Muto T, Bussey HJ, Morson BC. The evolution of cancer of the colon and rectum. Cancer. 1975 Dec;36(6):2251-70. doi: 10.1002/cncr.2820360944. PMID 1203876
- [Background] Vogelstein B, Fearon ER, Hamilton SR, Kern SE, Preisinger AC, Leppert M, Nakamura Y, White R, Smits AM, Bos JL. Genetic alterations during colorectal-tumor development. N Engl J Med. 1988 Sep 1;319(9):525-32. doi: 10.1056/NEJM198809013190901. PMID 2841597
- [Background] Winawer SJ, Zauber AG, Ho MN, O'Brien MJ, Gottlieb LS, Sternberg SS, Waye JD, Schapiro M, Bond JH, Panish JF, et al. Prevention of colorectal cancer by colonoscopic polypectomy. The National Polyp Study Workgroup. N Engl J Med. 1993 Dec 30;329(27):1977-81. doi: 10.1056/NEJM199312303292701. PMID 8247072
- [Background] Muller AD, Sonnenberg A. Prevention of colorectal cancer by flexible endoscopy and polypectomy. A case-control study of 32,702 veterans. Ann Intern Med. 1995 Dec 15;123(12):904-10. doi: 10.7326/0003-4819-123-12-199512150-00002. PMID 7486484
- [Background] Thiis-Evensen E, Hoff GS, Sauar J, Langmark F, Majak BM, Vatn MH. Population-based surveillance by colonoscopy: effect on the incidence of colorectal cancer. Telemark Polyp Study I. Scand J Gastroenterol. 1999 Apr;34(4):414-20. doi: 10.1080/003655299750026443. PMID 10365903
- [Background] Armitage N. Screening for cancer. In: Morris D, Kearsley, J, Williams, C, editor. Cancer: a comprehensive clnical guide. pp 9-20. U.K.: Taylor and Francis Ltd 1997.
- [Background] Mandel JS, Bond JH, Church TR, Snover DC, Bradley GM, Schuman LM, Ederer F. Reducing mortality from colorectal cancer by screening for fecal occult blood. Minnesota Colon Cancer Control Study. N Engl J Med. 1993 May 13;328(19):1365-71. doi: 10.1056/NEJM199305133281901. PMID 8474513
- [Background] Kronborg O, Fenger C, Olsen J, Jorgensen OD, Sondergaard O. Randomised study of screening for colorectal cancer with faecal-occult-blood test. Lancet. 1996 Nov 30;348(9040):1467-71. doi: 10.1016/S0140-6736(96)03430-7. PMID 8942774
- [Background] Hardcastle JD, Chamberlain JO, Robinson MH, Moss SM, Amar SS, Balfour TW, James PD, Mangham CM. Randomised controlled trial of faecal-occult-blood screening for colorectal cancer. Lancet. 1996 Nov 30;348(9040):1472-7. doi: 10.1016/S0140-6736(96)03386-7. PMID 8942775
- [Background] Lindholm E, Brevinge H, Haglind E. Survival benefit in a randomized clinical trial of faecal occult blood screening for colorectal cancer. Br J Surg. 2008 Aug;95(8):1029-36. doi: 10.1002/bjs.6136. PMID 18563785
- [Background] Atkin WS, Cook CF, Cuzick J, Edwards R, Northover JM, Wardle J; UK Flexible Sigmoidoscopy Screening Trial Investigators. Single flexible sigmoidoscopy screening to prevent colorectal cancer: baseline findings of a UK multicentre randomised trial. Lancet. 2002 Apr 13;359(9314):1291-300. doi: 10.1016/S0140-6736(02)08268-5. PMID 11965274
- [Background] Segnan N, Senore C, Andreoni B, Aste H, Bonelli L, Crosta C, Ferraris R, Gasperoni S, Penna A, Risio M, Rossini FP, Sciallero S, Zappa M, Atkin WS; SCORE Working Group--Italy. Baseline findings of the Italian multicenter randomized controlled trial of "once-only sigmoidoscopy"--SCORE. J Natl Cancer Inst. 2002 Dec 4;94(23):1763-72. doi: 10.1093/jnci/94.23.1763. PMID 12464648
- [Background] Schoen RE, Pinsky PF, Weissfeld JL, Yokochi LA, Church T, Laiyemo AO, Bresalier R, Andriole GL, Buys SS, Crawford ED, Fouad MN, Isaacs C, Johnson CC, Reding DJ, O'Brien B, Carrick DM, Wright P, Riley TL, Purdue MP, Izmirlian G, Kramer BS, Miller AB, Gohagan JK, Prorok PC, Berg CD; PLCO Project Team. Colorectal-cancer incidence and mortality with screening flexible sigmoidoscopy. N Engl J Med. 2012 Jun 21;366(25):2345-57. doi: 10.1056/NEJMoa1114635. Epub 2012 May 21. PMID 22612596
- [Background] Register of the total population: https://http://www.skatteverket.se/download/18.2b543913a42158acf80003761/1386594730871/Allm%C3%A4nBeskrivning.pdf: Swedish tax agency; [cited 2014 February].
- [Background] von Karsa L, Patnick J, Segnan N. European guidelines for quality assurance in colorectal cancer screening and diagnosis. First Edition--Executive summary. Endoscopy. 2012 Sep;44 Suppl 3:SE1-8. doi: 10.1055/s-0032-1309822. Epub 2012 Sep 25. PMID 23012113
- [Background] Rembacken B, Hassan C, Riemann JF, Chilton A, Rutter M, Dumonceau JM, Omar M, Ponchon T. Quality in screening colonoscopy: position statement of the European Society of Gastrointestinal Endoscopy (ESGE). Endoscopy. 2012 Oct;44(10):957-68. doi: 10.1055/s-0032-1325686. Epub 2012 Sep 17. No abstract available. PMID 22987217
- [Background] Patient register: http://www.socialstyrelsen.se/register/halsodataregister/patientregistret/inenglish: National Board of Health and Welfare; [cited 2014 February].
- [Background] Causes of Death register: http://www.socialstyrelsen.se/register/dodsorsaksregistret: National Board of Health and Welfare; [cited 2014 February].
- [Derived] Sekiguchi M, Westerberg M, Lowbeer C, Blom J, Forsberg A. First-Round Fecal Immunochemical Test Concentration Predicts Colorectal Cancer and Advanced Neoplasia in Second-Round Screening. Am J Gastroenterol. 2025 Aug 25. doi: 10.14309/ajg.0000000000003738. Online ahead of print. PMID 40853361
- [Derived] Westerberg M, Eriksson J, Metcalfe C, Lowbeer C, Ekbom A, Steele R, Holmberg L, Forsberg A. Colonoscopy findings after increasing two-stool faecal immunochemical test (FIT) cut-off: Cross-sectional analysis of the SCREESCO randomized trial. J Intern Med. 2024 Aug;296(2):187-199. doi: 10.1111/joim.13810. Epub 2024 Jun 6. PMID 38845164
- [Derived] Bonander C, Westerberg M, Chauca Strand G, Forsberg A, Stromberg U. Colorectal cancer screening with fecal immunochemical testing or primary colonoscopy: inequities in diagnostic yield. JNCI Cancer Spectr. 2024 Apr 30;8(3):pkae043. doi: 10.1093/jncics/pkae043. PMID 38830030
- [Derived] Westerberg M, Holmberg L, Ekbom A, Metcalfe C, Steele R, Forsberg A. The role of endoscopist adenoma detection rate in in sex differences in colonoscopy findings: cross-sectional analysis of the SCREESCO randomized controlled trial. Scand J Gastroenterol. 2024 Apr;59(4):503-511. doi: 10.1080/00365521.2023.2292480. Epub 2023 Dec 12. PMID 38084729
- [Derived] Sekiguchi M, Westerberg M, Ekbom A, Hultcrantz R, Forsberg A. Detection rates of colorectal neoplasia during colonoscopies and their associated factors in the SCREESCO study. J Gastroenterol Hepatol. 2022 Nov;37(11):2120-2130. doi: 10.1111/jgh.15990. Epub 2022 Sep 9. PMID 36062316
- [Derived] Stromberg U, Bonander C, Westerberg M, Levin LA, Metcalfe C, Steele R, Holmberg L, Forsberg A, Hultcrantz R. Colorectal cancer screening with fecal immunochemical testing or primary colonoscopy: An analysis of health equity based on a randomised trial. EClinicalMedicine. 2022 Apr 16;47:101398. doi: 10.1016/j.eclinm.2022.101398. eCollection 2022 May. PMID 35480071
- [Derived] Forsberg A, Westerberg M, Metcalfe C, Steele R, Blom J, Engstrand L, Fritzell K, Hellstrom M, Levin LA, Lowbeer C, Pischel A, Stromberg U, Tornberg S, Wengstrom Y, Ekbom A, Holmberg L, Hultcrantz R; SCREESCO investigators. Once-only colonoscopy or two rounds of faecal immunochemical testing 2 years apart for colorectal cancer screening (SCREESCO): preliminary report of a randomised controlled trial. Lancet Gastroenterol Hepatol. 2022 Jun;7(6):513-521. doi: 10.1016/S2468-1253(21)00473-8. Epub 2022 Mar 14. PMID 35298893
- [Derived] Shaukat A, Kahi CJ, Burke CA, Rabeneck L, Sauer BG, Rex DK. ACG Clinical Guidelines: Colorectal Cancer Screening 2021. Am J Gastroenterol. 2021 Mar 1;116(3):458-479. doi: 10.14309/ajg.0000000000001122. PMID 33657038
- [Derived] Wangmar J, von Vogelsang AC, Hultcrantz R, Fritzell K, Wengstrom Y, Jervaeus A. Are anxiety levels associated with the decision to participate in a Swedish colorectal cancer screening programme? A nationwide cross-sectional study. BMJ Open. 2018 Dec 22;8(12):e025109. doi: 10.1136/bmjopen-2018-025109. PMID 30580275

DOCUMENTS (2):
  • Study Protocol (2025-01-16): https://cdn.clinicaltrials.gov/large-docs/04/NCT02078804/Prot_002.pdf
  • Statistical Analysis Plan (2024-11-04): https://cdn.clinicaltrials.gov/large-docs/04/NCT02078804/SAP_001.pdf